CLINICAL TRIAL: NCT06683066
Title: Study on Human Bioequivalence of Triprerelin Acetate for Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Shandong Cancer Hospital and Institute (Other); Hunan Cancer Hospital (Other); Shanxi Province Cancer Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Chengdu Medical College (Other); Zibo Central Hospital (Other Government); Yuncheng Central Hospital (Other); Yichang Central People's Hospital (Other)
Responsible Party: Principal Investigator, Cao Yu, Director of the Phase I Clinical Research Center, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLG2051-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer (CRPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients must be in D - 28 hips intramuscular injection at a time Shot with acetic acid QuPu gonadorelin import (Diphereline) 3.75 mg, after screening the qualified with the method of delamination, block random, stratified factors for treatment (first time and the first) treatment, patients were randomly allocated to group A: T, Subjects were given triprelyn acetate for injection (manufactured and supplied by Qilu Pharmaceutical Co., LTD.) on the day of administration
  Interventions: Drug: Triprorelin for injection
- Group B (Active Comparator): All patients were injected 3.75mg triprerelin acetate (Diphereline) once into the buttock muscle of D-28 for introduction. After qualified screening, stratified and block randomized methods were adopted. Stratified factors were therapeutic factors (primary treatment and non-primary treatment), and patients were randomly assigned to group B :R, Subjects were given triprerelin acetate for injection on the day of administration (produced by Ipsen Pharma Biotech, supplied by Qilu Pharmaceutical Co., LTD.)
  Interventions: Drug: Diphereline

INTERVENTIONS:
Drug: Triprorelin for injection — Specification: Triprorelin for injection 3.75mg. Produced and supplied by Qilu Pharmaceutical Co.
  Arms: Group A
Drug: Diphereline — Specification: Diphereline 3.75mg. Produced by Ipsen Pharma Biotech and supplied by Qilu Pharmaceutical Co.
  Arms: Group B

SUMMARY:
To investigate the pharmacokinetics of triprerelin acetate for injection and triprerelin acetate (Dufferin ®) for injection of reference preparation in patients with prostate cancer by single intramusculodynamic injection in fasting state, and to evaluate the bioequivalence of the two formulations in fasting state.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the test, and sign the informed consent, and fully understand the test content, process and possible adverse reactions; 2. Male participants aged 18 years and older, male weight ≥50.0kg, body mass index (BMI) of 19 to 30kg/m2; 3. Patients with histopathologically diagnosed prostate cancer who were judged by investigators to be suitable for endocrine therapy, including 1 who had not received gonadotropin-releasing hormone analogues (GnRHa); 2 Patients receiving stable treatment with triprerelin acetate for injection; 3 Patients who have previously been treated with a gonadotropin-releasing hormone analogue (GnRHa) and who have been evaluated by the investigators as suitable for treatment with GNRHA; 4. ECOG score ≤2 points; 5. Expected survival ≥ 9 months; 6. Adequate hematopoietic function, liver and kidney function; 7. The subject is willing to have no family planning, sperm donation plan and voluntarily use one or more non-drug contraceptive methods (such as barrier contraception or abstinence) for 6 months from the signing of the information to the end of the drug administration.

-

Exclusion Criteria:

1. Patients who have previously undergone surgical castration; 2. Patients with known or suspected definite signs and symptoms of BMS or definite diagnosis of BMS; 3. Concurrent malignant tumors other than prostate cancer within 5 years, excluding basal cell carcinoma or squamous cell carcinoma of the skin that has been surgically removed; 4. Patients who have previously undergone adrenalectomy or pituitary resection or have pituitary disease; 5. Those who plan to undergo prostate surgery or other major surgical treatment during the study period (except urinary tract obstruction removal); 6. Patients with past or suspected spinal cord compression or urinary tract obstruction leading to kidney injury or patients at risk of developing such phenomena; 7. Patients with severe cardiovascular and cerebrovascular diseases, including but not limited to: patients with poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg under regular medication control); Patients with a history of hypertensive crisis or hypertensive encephalopathy; Severe cardiovascular and cerebrovascular disease, such as myocardial infarction, or heart failure classified by the New York Heart Association ≥II, within 6 months before the first administration of the investigational drug; Severe cardiac arrhythmia that cannot be controlled by medication (including QTc interval ≥470 ms), or congenital long QT syndrome; 8. Type I diabetes; Patients with type 2 diabetes with poor glycemic control (HbA1c>8.0% at screening); 9. Hepatitis B Surface antigen (HBsAg) test positive with HBV-DNA greater than 104copies/mL(or 2000IU/mL), or hepatitis C antibody positive with HCV-RNA test positive, or HIV antibody positive, Or syphilis antibody positive and RPR or TRUST positive; 10. Previous history of severe asthma or severe anaphylaxis or severe urticaria and/or vasogenic edema; 11. Persons known to be allergic to any component of triprerelin acetate for injection or to GnRH analogues; 12. People who are currently abusing drugs, drugs or alcohol (drinking an average of more than 14 units of alcohol per week, 1 unit =360 mL of beer or 45 mL of 40% alcohol spirits or 150 mL of wine); 13. A drug known to prolong the QT interval or induce tip torsive ventricular tachycardia (e.g., Class IA (e.g., quinidine, propylamine) or Class III (amiodarone, sotalol, dofetilide, ibutilide) was taken for 4 weeks or 5 half-lives (whichever is longer) prior to administration (including induction and trial) Psychotics, methadone, moxifloxacin, antipsychotics, etc; 14. Those who participate in other clinical trials and receive clinical trial drugs or devices within 1 month before administration (including the introduction period and the trial period); 15. Those who received any vaccine within 4 weeks prior to administration (including the introduction and trial period); 16. People who ingested special diet (such as grapefruit, pomelo and its products) within 48 hours before administration (including the introduction period and the trial period), or other factors that may affect drug absorption, distribution, metabolism, excretion and so on; 17. Those who donated blood or lost a large amount of blood (≥200mL) within 1 month before administration (including the introduction period and the trial period), and received blood transfusion or platelet transfusion ≥2 therapeutic amounts (1 therapeutic amount =12U platelet); 18. Patients with difficulty in venous blood collection; 19. Other circumstances in which the investigator considers it inappropriate to participate in the clinical trial, or in which the participant's participation in the trial may affect the trial results or his or her own safety.

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-04 (Estimated); Primary Completion 2025-09-04 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 672 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-28d) | 28 days
  Area under the drug concentration-time curve from time 0 to the 28d accurately measurable concentration at sample collection time
Area under the plasma concentration versus time curve (AUC7-28d) | 28 days
  Area under the drug concentration-time curve from time 7 to 28d accurately measurable concentration at sample collection time

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No